CLINICAL TRIAL: NCT04269122
Title: A Single-Center Study to Assess Plasma Ammonia Time-Normalized Area Under the Curve From Time Zero to 24 Hours and Rate of Ureagenesis in Healthy Adult Subjects
Brief Title: A Study to Assess Plasma Ammonia Time-Normalized Area Under the Curve and Rate of Ureagenesis in Healthy Adult Subjects
Status: Completed | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 301NHV01
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Ornithine Transcarbamylase Deficiency
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part 1: 30 eligible subjects will be asked to participate in 3 inpatient visits, each lasting up to 3 days (Day -1 to Day 2). Each visit will assess 24-hour ammonia levels in plasma and rate of urea production for 4 hours following ingestion of [1-13C]sodium acetate. Sodium acetate is used as a tracer to measure the rate of ureagenesis.
  Interventions: Other: No Intervention
- Part 2: 90 eligible subjects will be asked to participate in 1 inpatient visit, each lasting up to 3 days (Day -1 to Day 2). Each visit will assess 24-hour ammonia levels in plasma and rate of urea production for 4 hours following ingestion of [1-13C]sodium acetate. Sodium acetate is used as a tracer to measure the rate of ureagenesis.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention

SUMMARY:
The objective of the study is to characterize 24-hour plasma ammonia levels, characterize urea production rates in healthy normal subjects.

DETAILED DESCRIPTION:
During Part 1, eligible subjects will be asked to participate in 3 inpatient visits, each lasting up to 3 days (Day -1 to Day 2). Each visit will assess 24-hour ammonia levels in plasma and rate of urea production for 4 hours following ingestion of [1-13C]sodium acetate. Sodium acetate is used as a tracer to measure the rate of ureagenesis.

During Part 2, eligible subjects will be asked to participate in 1 inpatient visit, lasting up to 3 days (Day -1 to Day 2). The visit will assess 24-hour ammonia levels in plasma and rate of urea production for 4 hours following ingestion of [1-13C]sodium acetate. Sodium acetate is used as a tracer to measure the rate of ureagenesis.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 30 kg/m2, inclusive.

Exclusion Criteria:

* History of liver disease as evidenced by any of the following: portal hypertension, ascites, splenomegaly, esophageal varices, hepatic encephalopathy, or a liver biopsy with evidence of stage 3 fibrosis.
* Significant hepatic inflammation or cirrhosis as evidenced by imaging or any of the following laboratory abnormalities: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than the upper limit of normal (ULN), total bilirubin >1.5 × ULN, alkaline phosphatase >2.5 × ULN. NOTE: the ALT and/or AST levels may be repeated.
* Subject has a history of gout.
* Plasma ammonia level that is not within normal limits at Screening in the opinion of the Investigator or Sponsor.
* Received any vaccine within 14 days prior to Screening.
* Pregnant, lactating, or intending to become pregnant at any time during the study.
* Blood transfusion within 8 weeks prior to Screening.diuretics, cyclophosphamide and other cytotoxic agents, tolbutamide, chlorpropamide, diazoxide, dichlorphenamide, pyrazinamide, probenecid, theophylline/aminophylline, riluzole, warfarin and other antithrombotic agents, supplements containing aluminum hydroxide, or iron supplements within 30 days of Part 1or Part 2.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers at a Phase 1 unit
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Plasma Ammonia Area Under the Curve (AUC0-24) | Part 1, Day 1 (Visits 1-3) and Part 2, Day 1:Predose (0hour) up to 24 hours post dose
  Characterization of ammonia production over 24hr
Rate of Ureagenesis Based On Presence of [1-13C] In Urea | Part 1, Day 1 (Visits 1-3) and Part 2, Day 1: Predose (0hour) up to 4 hours post dose
  Characterization of nitrogen flux as determined by production of urea. Sodium acetate is used as a tracer to measure the rate of ureagenesis.
Intra- and inter-subject coefficient of variation (CV) of AUC0-24 and Rate of Ureagenesis | Part 1 Treatment Period: 17 days; Part 2 Treatment Period: 3 days
  Comparative analysis of both parameters

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical
Locations (1):
- PPD Phase 1 Unit, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No